CLINICAL TRIAL: NCT04869709
Title: Timing of Late Preterm Corticosteroid Administration and Neonatal Hypoglycemia
Brief Title: Late Preterm Corticosteroids and Neonatal Hypoglycemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Elizabeth Sasso, Assistant Professor of Obstetrics & Gynecology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APP-21-01310
Record Dates: First submitted 2021-04-09; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Neonatal Hypoglycemia; Prematurity
MeSH Terms: conditions — Premature Birth | interventions — betamethasone sodium phosphate; Betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Late Preterm Steroids 2 Days (Active Comparator)
  Interventions: Drug: Betamethasone Sodium Phosphate
- Late Preterm Steroids 7 Days (Active Comparator)
  Interventions: Drug: Betamethasone Sodium Phosphate

INTERVENTIONS:
Drug: Betamethasone Sodium Phosphate — Betamethasone Sodium Phosphate 12mg IM q24h for 2 doses
  Other Names: Celestone

SUMMARY:
This is a prospective randomized controlled trial investigating the timing of betamethasone administration in late preterm infants in relation to delivery and impact on neonatal hypoglycemia. Previous data has shown that neonatal hypoglycemia is increased in late preterm infants that were exposed to antenatal corticosteroids. The investigators hypothesize that the timing of steroid administration may impact the development of neonatal hypoglycemia.

DETAILED DESCRIPTION:
The use of antenatal corticosteroids for women at risk for preterm delivery has become widely adopted as standard of care. The American College of Obstetrics and Gynecologists (ACOG) officially recommends the use of corticosteroids for pregnant women between 24 and 34 weeks of gestation at risk of delivery within 7 days. Since publication of the ALPS trial, the Society of Maternal Fetal Medicine (SMFM) published guidelines supporting the use of late preterm steroids for singleton pregnancies between 34 weeks 0 days and 36 weeks 6 days who are at high risk of preterm birth within 7 days.

A secondary finding of the ALPS trial included the observation that the administration of antenatal betamethasone significantly increased the rate of neonatal hypoglycemia; the authors emphasized that while the long-term risks associated with neonatal hypoglycemia are not fully known, significant hypoglycemia is associated with poor neurodevelopmental outcome.

The optimal interval for administering late preterm steroids before delivery to minimize the risks of hypoglycemia while maximizing the benefits of fetal lung maturity has not been identified. The proposed research study will further investigate this question by randomizing patients to receive late preterm corticosteroids 2 days before delivery versus 7 days before delivery in order to determine if the rates and severity of neonatal hypoglycemia are different.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age 34 0/7 weeks to 36 5/7 weeks
* Planned delivery in late preterm period

Exclusion Criteria:

* Prior course of betamethasone during pregnancy
* Twin gestation
* Fetal demise
* Major fetal anomaly
* Maternal contraindication to betamethasone
* Pregestational diabetes
* Expected delivery within 12 hours of randomization

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Neonatal Glucose Concentration | Delivery to 72 hours of life
  Glucose reported in mg/dL; Hypoglycemia defined as concentration < 40 mg/dL

SECONDARY OUTCOMES:
Length of Hospital Stay | Delivery to discharge from hospital
  Days in hospital from date of delivery until date of discharge
Use of CPAP or High Flow Nasal Cannula | Delivery to 72 hours of life
  Drop in oxygen saturation requiring use of CPAP or high flow nasal cannula for at least 12 continuous hours
Need for supplemental oxygen | Delivery to 72 hours of life
  Drop in oxygen saturation requiring use of supplemental oxygen with a fraction of inspired oxygen (FiO2) of at least 0.30 for at least 24 continuous hours
Use of ECMO | Delivery to 72 hours of life
  Drop in oxygen saturation requiring use of ECMO (extracorporeal membrane oxygenation)
Use of mechanical ventilation | Delivery to 72 hours of life
  Drop in oxygen saturation and/or inability to maintain an airway requiring use of mechanical ventilation
Stillbirth | From administration of the intervention (betamethasone) to delivery
  Incidence of intrauterine fetal demise at any point after administration of the intervention (betamethasone) and before delivery
Neonatal death | Delivery to 30 days of life
  Death of fetus after delivery
Respiratory distress syndrome (RDS) | Delivery to 72 hours of life
  Defined as the presence of clinical signs of respiratory distress (ie: tachypnea, retractions, flaring, grunting, cyanosis) with a requirement of supplemental oxygen with a fraction of inspired oxygen of more than 0.21 and a chest radiograph showing hypoaeration and reticulogranular infiltrates
Transient Tachypnea of the Newborn | Delivery to 72 hours of life
  Defined when tachypnea (Respiratory Rate >60 breaths per minute) occurs in the absence of chest radiography or a radiograph that was normal and resolved within 72 hours
Need for surfactant administration | Delivery to 72 hours of life
  Need for administration of exogenous surfactant in the setting of neonatal respiratory distress
Neonatal pneumonia | Delivery to 72 hours of life
  Defined when a combination of clinical, microbiologic, and/or radiographic findings suggest primary pulmonary infection as a cause of respiratory distress, fevers, increasing white blood cell count, need for antibiotics, and/or sepsis.

OTHER OUTCOMES:
Need for resuscitation at birth | Within 30 minutes of delivery
  Any intervention in the first 30 minutes, excluding blow-by oxygen
Neonatal Hypothermia | Delivery to 72 hours of life
  Defined as rectal temperature below 36 degrees Celsius
Necrotizing Entercolitis | Delivery to 72 hours of life
  When systemic, radiographic, and abdominal signs lead to a modified Bell stage 2 or 3
Intraventricular Hemorrhage Grade 3 or 4 (Severe IVH) | Delivery to 72 hours of life
  Defined when the extent of brain injury includes a hemorrhage that occupies more than 50% of the lateral ventricle volume
Feeding Difficulty | Delivery to 72 hours of life
  inability to take all feeds by mouth, requiring gavage feeds or intravenous supplementation at least once.

CONTACTS AND LOCATIONS:
Locations (1):
- LAC+USC Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Practice Bulletin No. 159: Management of Preterm Labor. Obstet Gynecol. 2016 Jan;127(1):e29-e38. doi: 10.1097/AOG.0000000000001265. PMID 26695585
- [Background] Liggins GC, Howie RN. A controlled trial of antepartum glucocorticoid treatment for prevention of the respiratory distress syndrome in premature infants. Pediatrics. 1972 Oct;50(4):515-25. No abstract available. PMID 4561295
- [Background] Gyamfi-Bannerman C, Thom EA, Blackwell SC, Tita AT, Reddy UM, Saade GR, Rouse DJ, McKenna DS, Clark EA, Thorp JM Jr, Chien EK, Peaceman AM, Gibbs RS, Swamy GK, Norton ME, Casey BM, Caritis SN, Tolosa JE, Sorokin Y, VanDorsten JP, Jain L; NICHD Maternal-Fetal Medicine Units Network. Antenatal Betamethasone for Women at Risk for Late Preterm Delivery. N Engl J Med. 2016 Apr 7;374(14):1311-20. doi: 10.1056/NEJMoa1516783. Epub 2016 Feb 4. PMID 26842679
- [Background] Society for Maternal-Fetal Medicine (SMFM) Publications Committee. Implementation of the use of antenatal corticosteroids in the late preterm birth period in women at risk for preterm delivery. Am J Obstet Gynecol. 2016 Aug;215(2):B13-5. doi: 10.1016/j.ajog.2016.03.013. Epub 2016 Mar 15. No abstract available. PMID 26992737
- [Background] Kamath-Rayne BD, Rozance PJ, Goldenberg RL, Jobe AH. Antenatal corticosteroids beyond 34 weeks gestation: What do we do now? Am J Obstet Gynecol. 2016 Oct;215(4):423-30. doi: 10.1016/j.ajog.2016.06.023. Epub 2016 Jun 21. PMID 27342043
- [Background] Uquillas KR, Lee RH, Sardesai S, Chen E, Ihenacho U, Cortessis VK, Barton L. Neonatal hypoglycemia after initiation of late preterm antenatal corticosteroids. J Perinatol. 2020 Sep;40(9):1339-1348. doi: 10.1038/s41372-020-0589-1. Epub 2020 Feb 14. PMID 32060360